CLINICAL TRIAL: NCT04458636
Title: Delivering Personalised Care in the Management of Exacerbations of Chronic Obstructive Pulmonary Disease: A Multi-centre Randomised Clinical Trial
Brief Title: Stratified TreAtment to Reduce Risk in COPD
Acronym: STARR2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Mona Bafadhel, Associate Professor, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17/LO/1135
Record Dates: First submitted 2017-08-20; First posted 2020-07-07 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: COPD Exacerbation
Keywords: eosinophils; oral corticosteroids; primary care
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Blinded prednisolone 30mg orally once per day for 14 days
  Interventions: Drug: Prednisolone
- Biomarker care (Placebo Comparator): Blinded prednisolone 30mg orally once per day for 14 days if peripheral eosinophil count is equal or greater than 2%. Placebo equivalent if peripheral blood eosinophil count is <2%.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Oral

SUMMARY:
To evaluate the efficacy of blood-eosinophil directed corticosteroid therapy using near-patient testing, compared to current standard practice during an exacerbation of COPD in a multi-centre randomised placebo controlled trial.

DETAILED DESCRIPTION:
Study design: Double-blind placebo controlled randomised clinical trial Study setting: Primary care GP practices Participants: Adults ≥40 years with COPD Sample size: 228 Study duration: 12 months data collection Primary objective: To evaluate the efficacy of blood-eosinophil directed corticosteroid therapy using near-patient testing, compared to current standard practice during an exacerbation of COPD.

Secondary objective: To evaluate quality of life, symptoms, lung function and healthcare utilisation in a blood-eosinophil directed corticosteroid therapy arm.

Exploratory objective: To evaluate stability of eosinophil counts and mediator levels

Chronic obstructive pulmonary disease (COPD) affects adults and is largely caused by cigarette smoke in the developed world. It is predicted to be the 3rd leading cause of death by 2020 affecting over 250 million people worldwide. COPD is characterised by progressive airflow obstruction punctuated by frequent periods of worsening in respiratory symptoms and function associated with a significant impact on quality of life. These episodes are termed exacerbations and current treatment strategies rely on oral corticosteroids (prednisolone) and antibiotics but this is in a "one size fits all" approach. However there is little evidence supporting this strategy and both treatments can potentially cause harm. In addition to this, previous findings have shown that eosinophil counts within blood samples from COPD patients can be used as a biomarker to determine treatment with oral steroids.

The use of near-patient testing in primary care will characterise patients with COPD and inform to guide effective and personalised treatment with reductions in treatment failure rates, improvements in health and reductions in adverse events associated with inappropriate and excessive corticosteroid and antibiotic therapy. Currently available systems include the HemoCue ® 5-point differential cell count system which accurately and rapidly (within 2 minutes) determine the eosinophil count finger-prick sampling. This diagnostic is currently used in neonatology, Emergency Departments (ED) and at Mount Everest Base Camp 28-30. It is thus conceivable that this could be used in primary care to deliver a randomised control trial to demonstrate that stratified medicine approaches in the management of COPD exacerbations are superior to standard therapy.

It is believed that personalising this treatment approach during an exacerbation of COPD, to direct whether corticosteroids is necessary for all patients, depending on the results of the eosinophil count from near-patient testing, is superior to current standard treatment strategies in the primary care setting.

Recruitment target for STARR 2 is 228 participants with COPD from GP surgeries within the Thames Valley and South Midlands. A participant's involvement is 12 months and involves up to 5 visits. These visits consist of CRF completion, questionnaires, breathing tests, urine testing, blood samples and spirometry. The trial drugs are only taken for 14 days during an exacerbation but participants can be re-randomised for up to 4 times in the study when they exacerbate.

Intervention: At exacerbation randomised to 'standard therapy' or 'blood eosinophil directed therapy'. Standard therapy will be prednisolone and antibiotic therapy. Blood eosinophil directed therapy will be prednisolone and/or antibiotic therapy.

Investigational medicinal product: Prednisolone or placebo equivalent. The IMP is part of current clinical practice. Prednisolone is an anti-inflammatory and given in short durations (≤2 weeks duration) orally for its systemic action at the onset of an exacerbation in COPD.

Participation duration: Study entry at stable state or during an exacerbation. Randomisation at exacerbation. IMP treatment period 14 days. Post treatment follow-up visits at days 14, 30 and 90. Stable state and randomisation visit duration maximum 60 minutes. Follow-up visits at days 14, 30, and 90 maximum duration 30 minutes. Participants may be re-randomised and followed up if they have further exacerbations after the 30 day visit.

Data collection: Demographic and exacerbation clinical data including duration of symptoms, past medical history, medication history and exacerbation history is collected. Blood eosinophil tests is collected by pin-prick testing using the HemoCue ®; lung function using spirometry and FeNO; and symptoms and quality of life using questionnaires. Serum is collected at visits.

Study schedule:

Study assessments will be performed within primary care by the research study team. The following assessments may occur at the study visits:

Eligibility check: Inclusion and exclusion criteria will be checked against the participant's medical notes and with the participant during the visit. This responsibility will be delegated by the PI to a member of the research team.

Demographic history: Participant demographics including age, smoking history and past COPD medical history will be collected.

Medication history: Full medication history will be collected, including the use of as required and over the counter medication. Any drug allergy will be documented and dates of flu vaccination, S. pneumoniae and H. influenzae B vaccinations will be recorded from medical records.

Past medical history: Full medical history will be collected from the participant and from the medical notes. COPD diagnosis history: The age of onset and age of diagnosis of COPD symptoms will be recorded from the participant and from the medical records.

Past exacerbation history: The frequency of exacerbations, including those requiring hospitalisation in the previous 12 months will be captured from participant recollection and from the medical records. Medication prescribed at each exacerbation event (if available) from medical records will be captured.

Exacerbation history: The current history of the exacerbation, including duration of symptoms and treatment history will collected by questioning. The severity of the exacerbation will be recorded according to Anthonisen criteria14 with increased symptoms of breathlessness, sputum production and sputum purulence will be used as per GOLD31 definition. The Anthonisen criteria for exacerbation as follows: Type 1 - Three major symptoms; Type 2 - two major symptoms; Type 3 - One major and one minor symptom. The major symptoms are i) Increased breathlessness; ii) increased sputum production; or iii) increased sputum purulence. The minor symptoms are iv) Upper respiratory tract infection in the previous 5 days; v) fever without apparent cause; vi) increased wheeze; vii) increased cough; viii) increase in respiratory or heart rate 20% above baseline. Questionnaires: Patient reported outcome measures (PRO's) will be sought to specifically test symptoms, health status, quality of life and any associated depression and anxiety. This will include the Medical Research Council dyspnoea scale (MRC); Visual analogue score (VAS) 32; COPD Assessment Tool (CAT) 33; the Hospital Anxiety and Depression Scale (HADS)34 and the EuroQol 5D35. Participants will be asked to complete a daily diary (using the VAS tool, for the duration of 30 days) for assessment of symptoms and recovery following treatment. Instructions to use these questionnaires will be given to all participants. Each of these questionnaires are validated to be self-completed for ease of use. All research staff undertaking any assessments and procedures will be trained to use the equipment and perform the questionnaires to determine patient reported outcomes. Near-patient point of care testing procedures:

Approximately 5 drops of blood (up to a maximum of 10 drops) will be taken for measurement of peripheral blood eosinophil counts, glucose and CRP levels.

A urine sample for testing of glycosuria will be performed immediately. All samples will be discarded.

Lung Function: Spirometry will be performed to determine the forced expiratory volume in 1 second (FEV1) and the forced vital capacity (FVC) according to standard ATS/ERS criteria36.

Venous blood sampling: Using a fully sterile technique, a blood test will be performed to measure inflammation. All participants consenting to trial sample collection will have a maximum of 20mLs of blood taken at each visit. Collected blood will be centrifuged immediately and serum/plasma will be aliquoted into fully anonymised barcoded tubes. Anonymised samples will be then be securely transported to the John Radcliffe Hospital and stored at the Respiratory Medicine Laboratory (John Radcliffe Hospital), under the HTA licence, at -80˚c for exploratory outcome analysis and for future use subject to ethical approval. There will be separate instructions detailing the sample handling process for this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 40 years or above.
* Diagnosed with COPD (primary or secondary care diagnosis) with spirometric confirmation of airflow obstruction (FEV1/FVC ratio <0.7).
* A history of at least 1 exacerbation in the previous 12 months, requiring systemic corticosteroids and/or antibiotics.
* Current or ex-smoker with at least a 10 pack year smoking history
* In the opinion of the research staff, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* History of atopic childhood asthma
* Current history of primary lung malignancy or current active pulmonary TB
* Clinically relevant disease or disorder (past or present) which in the opinion of the investigator may either put the subject at risk because of participating in the study or may influence the results of the study or the subject's ability to participate in the study.
* Any clinically relevant lung disease, other than COPD considered by the investigator to be the primary diagnosis. For example mild-to-moderate bronchiectasis is acceptable in addition to COPD unless the bronchiectasis is considered to be the primary diagnosis.
* An alternative cause for the increase in symptoms of COPD that are unrelated to an exacerbation such as i) suspicion or clinical evidence of pneumonia; ii) high probability and suspicion of pulmonary embolism; iii) suspicion or clinical evidence of a pneumothorax; iv) primary ischaemic event - ST or Non ST elevation myocardial infarct and left ventricular failure [i.e. not an exacerbation of COPD]
* A known allergy to the IMP (prednisolone), NIMP (doxycycline) or to any of the constituents of the placebo
* Patients on maintenance corticosteroids (prednisolone, hydrocortisone, fludrocortisone)
* Known adrenal insufficiency
* Currently enrolled in another CTIMP trial and receiving an intervention as part of the trial.
* Pregnant and breast-feeding women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of treatment non-responders defined as those needing re-treatment, hospitalisation or death at 30 and 90 days | 30 days
  Frequency of treatment non-responders, defined as those needing re-treatment, hospitalisation or death

SECONDARY OUTCOMES:
COPD assessment test (CAT) | Day 14, 30 and 90
  CAT questionnaire. A higher score (max score of 40) reflects worse COPD symptoms
Quality of life - change from baseline | Day 14, 30 and 90
  European Quality of Life-5 dimension-3 level (EQ 5D 3L) questionnaire. A higher number on each of the 5 dimension reflects worse quality of life
Visual analogue scale (VAS) for cough, wheeze, sputum volume, sputum purulence and breathlessness | Day 14, 30 and 90
  Visual Analogue Scale (VAS) symptom score (scale of 0 to 100 - 100 being the worst). Separate scale for 5 items: cough, wheeze, sputum volume, sputum purulence and breathlessness. Results will be represented as a sum of all 5 scores at each time point.
Lung function | Day 14, 30 and 90
  Change from baseline in FEV1
Exacerbations | 12 months
  Frequency of moderate and severe exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bafadhel, MBChB, PhD, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Department of Medicine, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
upon request

REFERENCES:
- See also: Website address for CI — https://www.ndm.ox.ac.uk/principal-investigators/researcher/mona-bafadhel